CLINICAL TRIAL: NCT06457360
Title: Comparative Assessment of Chitosan-Based Dressing, Ankaferd and Tranexamic Acid in Achieving Hemostasis and Healing Following Dental Extraction in Liver Pre-Transplant Children
Brief Title: Comparison of Chitosan, Ankaferd and Tranexamic Acid in Dental Extraction in Liver Pre-Transplant Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PED 20-2D
Record Dates: First submitted 2023-11-22; First posted 2024-06-13 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Tranexamic Acid; ankaferd blood stopper; Chitosan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 sterile gauze with chitosan (Experimental): Chitosan-based dressing gauze after extraction in patients with end stage liver disease
  Interventions: Drug: Chitosan
- group 2 sterile gauze with ankaferd blood stopper (Experimental): ankaferd blood stopper dressing gauze after extraction in patients with end stage liver disease
  Interventions: Drug: Ankaferd Blood Stopper
- group 3 sterile gauze with tranexamic acid (Active Comparator): tranexamic acid dressing gauze after extraction in patients with end stage liver disease
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — Application of sterile gauze after extraction for hemostasis
  Arms: group 3 sterile gauze with tranexamic acid
Drug: Ankaferd Blood Stopper — Application of sterile gauze after extraction for hemostasis
  Arms: group 2 sterile gauze with ankaferd blood stopper
Drug: Chitosan — Application of sterile gauze after extraction for hemostasis
  Arms: group 1 sterile gauze with chitosan

SUMMARY:
The aim of the present study is:

To assess the hemostatic effect of chitosan-based dressing, Ankaferd and Tranexamic acid after extraction in children with end stage liver diseases where the:

• Primary objective: is to evaluate which of the previous materials will be the most effective as a hemostatic agent

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end stage liver disease that need dental extraction before liver transplant
2. Patients aged between 4 and 9 years old
3. Patients having international normalized ratio (INR) values ≤ 4 (i.e. 1-4)

Exclusion Criteria:

1. Patients with allergy to sea food because chitosan- based dressing is manufactured from freeze-dried chitosan, derived from shrimp shell.
2. Patients having genetic bleeding disorders
3. Patients with renal diseases

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
To assess the hemostatic effect of chitosan-based dressing, Ankaferd and Tranexamic acid after extraction in children with end stage liver diseases | 30 minutes
  evaluation of the previous materials which will be the most effective as a hemostatic agent by measuring blood loss after dental extraction after 30 minutes by the weight difference between the gauze preoperatively and postoperatively using fine electronic measurement weight device

SECONDARY OUTCOMES:
pain score assessment | 7 days
  Pain scores will be assessed using Visual Analog Scale from 0 to 10 pain score for seven days following extraction where 0 is no pain and 10 is maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: noha S Kabil, Principal Investigator — British University In Egypt
Locations (1):
- British University in Egypt, Cairo, Egypt